CLINICAL TRIAL: NCT03740776
Title: The Eosinophils Percentage Predicts In-hospital Major Adverse Cardiac Events in Patients With ST-elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention
Brief Title: The Eosinophils Percentage Predicts In-hospital Major Adverse Cardiac Events in STEMI Patients After PCI
Status: Completed | Type: Observational
Sponsor: Dongying Zhang (Other)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Professor, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 2018-35
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophils (EOS) in peripheral blood are significantly decreased in ST-segment elevation myocardial infarction (STEMI) and the reduced EOS indicates severe myocardial damage. Whether EOS is a good predictor for in-hospital major adverse cardiac events (MACEs) of patients with ST-segment elevation myocardial infarction remains unknown. The aims of this study was to evaluate prognostic role of EOS for in-hospital MACEs in STEMI patients who have undergone primary percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
The investigators retrospectively analyzed the clinical data of 518 patients with STEMI after PCI. MACEs were defined as cardiac arrest, cardiac rapture, malignant arrhythmia and cardiac death. The receiver operating characteristic (ROC) curves were used to demonstrate the prognostic value of EOS% in in-hospital MACEs. All patients were divided into 2 groups according to the best cut-off EOS% value, including reduced EOS% group and control group. Cox regression analyses and KM survival curve were used to calculate the correlated between EOS with in-hospital MACEs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI who underwent PCI within 12 hours from symptom onset
2. Patients from whom informed consent has been properly obtained in writing prior to start of the trial.

Exclusion Criteria:

1. Patients with previous myocardial infarction, congenital heart disease
2. Patients with liver disease, and renal failure
3. Patients with immunologic disease, malignant tumors, pregnancy, infection caused by various pathogens, chronic inflammatory disease, trauma.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: STEMI Patients
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events | The median time of 7 days
  the relationship between reduced eosinophils percentage and in-hospital MACE

IPD SHARING:
Plan to Share IPD: Undecided